CLINICAL TRIAL: NCT01237925
Title: Non-inferiority, Monocentric Comparative Open Study of Two Topical Pharmaceutical Preparations (Cream and Gel) of Dexchlorpheniramine Maleate in the Evaluation of Safety and Efficacy for the Relief of Mild to Moderate Sunburn Related Symptoms
Brief Title: Non-inferiority Clinical Trial of Dexchlorpheniramine (Cream Versus Gel) in the Relief of Sunburn Related Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Mantecorp Industria Quimica e Farmaceutica Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERE 185v2-10
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Sunburn
Keywords: Sunburn; Dexchlorpheniramine; Gel; Cream
MeSH Terms: conditions — Sunburn | interventions — dexchlorpheniramine; Gels

ARMS (2):
- Dexchlorpheniramine 1% gel (Experimental)
  Interventions: Drug: Dexchlorpheniramine 1% gel
- Dexchlorpheniramine 1% cream (Active Comparator)
  Interventions: Drug: Dexchlorpheniramine 1% cream

INTERVENTIONS:
Drug: Dexchlorpheniramine 1% gel — Small amount applied over the lesion twice a day for 7 days
  Arms: Dexchlorpheniramine 1% gel
Drug: Dexchlorpheniramine 1% cream — Small amount applied over the lesion twice a day for 7 days
  Arms: Dexchlorpheniramine 1% cream

SUMMARY:
Topical antihistamines can be used to promote relief of sunburn related symptoms (erythema, itch and burning sensations). Dexchlorpheniramine maleate 1% cream is a topical antihistamine formulation approved by ANVISA in Brazil for the relief of skin irritation and pruritus, including the ones caused by sunburn. The aim of the present study is to demonstrate non-inferiority of a new pharmacological preparation of dexchlorpheniramine maleate (1% gel) with the standard preparation (1% cream) for the relief of sunburn related symptoms and to demonstrate the safety of both preparations.

ELIGIBILITY:
Inclusion Criteria:

* Signs of solar erythema of mild to moderate intensity resulting from voluntary exposure to sun within the last 72 hours
* Compliance of the subject to the treatment protocol
* Agreement with the terms of the informed consent by the participants or their legal guardians when younger than 18 years old

Exclusion Criteria:

* Pregnancy or risk of pregnancy
* Lactation
* Signs of severe sunburn (vesicles, bullae or ulceration)
* Use of topical or systemic anti-inflammatory, antihistamine or immunosuppressive drugs within the last 48 hours prior to the study
* History of atopy or allergic diseases
* History of allergy to any component of the formulations
* Other conditions considered by the investigator as reasonable for non-eligibility

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)

PRIMARY OUTCOMES:
Pruritus intensity evaluated with a 10-point Visual Analogic Scale (VAS) | 7 days
  The evaluation of the pruritus will be made by a 10-point visual analog scale, answered by patients at each visit. The sum of weighted scores will be calculated for each sign / symptom in each patient.

SECONDARY OUTCOMES:
Composite clinical evaluation of erythema, pruritus and burning sensation performed by the investigator using a 4-point scale for each one of the variables (absent, mild, moderate, intense). | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda, Osasco, São Paulo, Brazil